CLINICAL TRIAL: NCT00334100
Title: Treadmill Training in Chronic MS: Efficacy and Cost-Effectiveness
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruiting
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3603-P; B3603-P (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; multiple sclerosis; treadmill
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Treadmill exercise

SUMMARY:
The purpose of the study is to determine whether treadmill training is safe and beneficial in patients with walking difficulty because of multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic inflammatory demyelinating disease of the central nervous system, which can cause episodic, static or progressive disability. Frequently, MS causes weakness and spasticity of the legs leading to gait abnormalities and immobility. Rehabilitation has been widely used in MS but has been the subject of limited investigation. In particular, traditional thinking in MS providers was that aerobic exercise could cause worsening of symptoms in some patients and should generally be avoided. Recent studies suggest that both aerobic exercise is tolerated by most patients and improves fitness. In a recent study however, training with bicycle ergometers did not translate into improved biomechanics of gait. This suggests that aerobic training may need to be coupled to task specific training to produce improved gait. With recent changes in medical care focusing on cost containment, studies supporting the effectiveness and cost-effectiveness of rehabilitation interventions are needed.

Studies from the stroke literature suggest that task specific training may be useful in promoting motor reorganization in the cortex, reversing muscle wasting and improving cardiovascular de-conditioning. In particular, we have examined the use of treadmill training in patients with chronic hemiparesis due to stroke and have found that a course of training can improve walking ability, can cause an increase in motor representation of the effected limb as measured by fMRI, can increase muscle mass as measured by thigh CT and muscle biopsy, and can improve cardiovascular fitness as measured by treadmill stress testing.

Proposed is a pilot study testing a program of treadmill training in patients with chronic leg weakness and spasticity due to MS causing chronic gait problems. The primary objectives of this pilot study are to demonstrate the safety and tolerability of the treadmill training program in MS patients and to obtain preliminary data on outcomes to use to determine the sample size for a larger trial designed to document efficacy and cost-effectiveness. Forty MS patients with impaired ambulation will be randomized to a 3 month program of treadmill training or a 3 month education and counseling program with attention equal to the treadmill trained group. Both groups will be followed for a total of 6 months. The treadmill training will be carried out in the Senior Exercise Research Center at the Baltimore VAMC. Outcome measures will include measures of leg strength and spasticity, disability (EDSS), walking ability, cardiovascular fitness, Quality of Life, depression, and healthcare costs and utilization (compared to the year prior to enrollment). The results of this pilot study will be used to design and gain support for a study sized to measure efficacy and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Chronic definite multiple sclerosis
* Visible paraparetic gait deficits
* EDSS 4 to 6.5
* Last 12 months of care in VHS
* Competent to provide consent and carry out study procedures
* Pass the Functional Mobility Entry Test

Exclusion Criteria:

* Performing 20 minutes or more of aerobic exercise 3X per week
* Alcohol consumption over 2 oz liquor, 8 oz wine, 24 oz beer per day
* Cardiac history
* Significant medical history
* Significant neurological history
* Relapsing MS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Primary Completion 2011-09 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 Treadmill, Step activity monitors, Timed 8 meter walk | Pre study and 12 weeks Post study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bever, MD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States